CLINICAL TRIAL: NCT05640609
Title: A Phase Ib/II Trial of Capeox Regimen Combined With Sintilimab and Bevacizumab in First-line Treatment for Recurrent or Metastatic Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Capeox Regimen Combined With Sintilimab and Bevacizumab for Gastric Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ming Liu, Associate Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 250260270
Record Dates: First submitted 2022-11-13; First posted 2022-12-07 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capeox regimen combined with Sintilimab and Bevacizumab (Experimental): Capeox regimen combined with Sintilimab and Bevacizumab
  Interventions: Combination Product: Capeox regimen combined with Sintilimab and Bevacizumab

INTERVENTIONS:
Combination Product: Capeox regimen combined with Sintilimab and Bevacizumab — Stage Ib：Oxaliplatin +Capecitabine Tablets +Sintilimab +Bevacizumab Stage II：Bevacizumab (the dose determined in phase Ib clinical study)，the dosage of other drugs was the same as before

SUMMARY:
The median survival time of first-line chemotherapy for advanced gastric cancer is about one year, and the treatment is still facing the bottleneck. This is a one-arm, open and prospective phase II clinical study. Recruit patients who have been diagnosed with advanced or metastatic adenocarcinoma of the stomach and gastroesophageal junction and have not received systematic treatment.

DETAILED DESCRIPTION:
The median survival time of first-line chemotherapy for advanced gastric cancer is about one year, and the treatment is still facing the bottleneck. Bevacizumab is an anti-vascular endothelial growth factor (VEGF) targeted therapy drug. It is doubtful whether the low dose of bevacizumab in gastric cancer patients leads to poor curative effect. Now the treatment of advanced gastric cancer has come to the era of immunotherapy. The chemotherapy regimen of daclizumab combined with CAPEOX has been proved to be effective in clinical studies. No clinical study has confirmed the safety and efficacy of CAPEOX regimen combined with sintilimab and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis confirmed adenocarcinoma of stomach and gastroesophageal junction (including signet ring cell carcinoma, mucinous adenocarcinoma, hepatoid adenocarcinoma)
2. Imaging and surgical evaluation of unresectable recurrent or metastatic patients
3. The expected survival time was more than 3 months
4. The age is between 18 and 70 years old, both male and female
5. No systematic treatment has been given to patients with advanced or metastatic gastric and esophagogastric junction adenocarcinoma.If the patients who have received adjuvant or neoadjuvant therapy (including chemotherapy, radiotherapy and chemotherapy), the last treatment must be completed at least 6 months before randomization, and there is no recurrence or disease progression at the time of treatment.Palliative radiotherapy was allowed, but it must be completed at least 2 weeks before the first study treatment.Subjects were allowed to receive anti-tumor traditional Chinese medicine preparations in the past, but they must be discontinued at least 2 weeks before randomization
6. Eastern Cooperative Oncology Group(ECoG) - 1 physical status
7. At least one lesion can be evaluated according to RECIST 1.1 criteria
8. It can provide pathological tissues or fresh pathological tissues that are filed within 6 months after the signature of informed consent for screening, and can obtain the test results. For the slices filed within 6 months before randomization, it should be confirmed that no systematic treatment (including adjuvant / neoadjuvant therapy) has been received after obtaining the samples
9. The function of the main organs is normal, that is to say, it meets the following standards:

   1. Blood routine examination (no blood transfusion within 14 days before screening)
   2. Hemoglobin ≥ 90 g / L;
   3. Absolute neutrophil count (ANC) ≥ 1.5×109/L;
   4. Platelet count ≥ 75×109/L; Blood biochemical test (albumin was not used within 14 days before screening)
   5. Albumin ≥ 28 g / L;
   6. Total bilirubin ≤ 1.5×Upper limit of normal value (ULN);
   7. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3×ULN; If there is liver metastasis, aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 5×ULN
   8. Creatinine ≤ 1.5×ULN;Coagulation function:
   9. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5×ULN;
   10. Activated partial thromboplastin time (APTT) ≤ 1.5×ULN
10. For sections filed in the first 6 months of randomization, it should be confirmed that no systematic treatment (including adjuvant / neoadjuvant therapy) has been received since sample acquisition
11. Acute toxicity caused by previous anti-tumor treatment or surgery was relieved to grade 0-1 (according to ncictcae 5.0) or to the level specified in the inclusion / exclusion criteria
12. Female subjects of childbearing age were required to conduct a serum pregnancy test within 3 days before the start of the study, and the results were negative, and they were willing to use a medically recognized high-efficiency contraceptive method (such as intrauterine device, contraceptive or condom) during the study period and within 3 months after the last administration of the study drug;For male subjects whose partners are women of childbearing age, they should be sterilized by surgery or agree to use effective contraceptive methods during the study and within 3 months after the last study administration
13. With my consent and signed the letter of understanding, I am willing and able to follow the planned visit, research treatment, laboratory examination and other test procedures

Exclusion Criteria:

1. HER2 + (or HER2 +) is known to be positive
2. Gastric cancer known as squamous cell carcinoma, undifferentiated or other tissue types, or adenocarcinoma mixed with other tissue types
3. There are uncontrolled or symptomatic active central nervous system (CNS) metastases, which can be characterized by clinical symptoms, brain edema, spinal cord compression, cancer metastasis, malignant meningitis, leptomeningeal disease, and / or progressive growth.Patients with CNS metastases can be enrolled in the study if they are adequately treated and their psychiatric symptoms can return to baseline level at least 2 weeks before randomization (except for residual signs or symptoms related to CNS treatment).In addition, subjects were required to discontinue corticosteroids or receive prednisone (or equivalent other corticosteroids) at least 2 weeks before randomization, or to receive a stable or gradually reduced dose of prednisone (or equivalent) at least 2 weeks before randomization
4. There were hydrothorax and ascites which could not be controlled by puncture and drainage within 14 days before the random;Pericardial effusion with clinical symptoms or moderate or above
5. The weight of the subjects decreased by more than 20% in the first two months of randomization
6. The following treatments or drugs were received before randomization: a) major surgery was performed within 28 days before randomization (tissue biopsy and peripherally inserted central catheter operation peripherally inserted central venous catheter （PICC） for diagnosis are allowed; b) immunosuppressive drugs were used within 7 days before randomization,Does not include nasal and inhaled corticosteroids or physiological doses of systemic hormones (i.e. no more than 10 mg / D of nisone or other corticosteroids with equivalent physiologic doses);c) Live attenuated vaccine was administered within 28 days before randomization or within 60 days after the end of drug treatment;d) Antineoplastic therapy (including chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, biotherapy or tumor embolization) within 28 days before randomization
7. Any other malignant tumor was diagnosed within 3 years before entering the study, except basal cell carcinoma of skin or squamous or superficial bladder cancer, carcinoma in situ of cervix, intraductal carcinoma of breast and papillary thyroid carcinoma that can be treated locally and cured.
8. There is any active, known or suspected autoimmune disease.Subjects who were in a stable state and did not need systemic immunosuppressive therapy were allowed to be included, such as type I diabetes mellitus, hypothyroid diabetes mellitus requiring hormone replacement therapy only, and skin diseases without systemic treatment (e.g., vitiligo, psoriasis and alopecia)
9. Previously received anti-PD-1 / PD-L1 antibody, anti-CTLA-4 antibody or other drugs acting on T-cell co stimulation or examination cell co stimulation or checkpoint pathway
10. There were significant bleeding symptoms or bleeding tendency in 3 months before random;Gastrointestinal perforation and / or gastrointestinal fistula occurred within 6 months before randomization;Arteriovenous thrombosis events occurred in the first 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc
11. Major vascular disease (e.g. aortic aneurysm requiring surgical repair or recent peripheral artery thrombosis) within 6 months before the start of study treatment
12. Severe, unhealed or dehiscent wounds and active ulcers or untreated fractures
13. There were peripheral neuropathy > 1 grade
14. If the symptoms of ileus (ileus) at the beginning of the study (with or without complete parenteral nutrition treatment) and symptoms of ileus were resolved at the time of initial diagnosis or complete parenteral nutrition treatment, or if the patient did not have the symptoms of ileus at the time of initial diagnosis / treatment, or had not received complete parenteral nutrition treatment,Patients may be admitted to the study
15. Interstitial lung disease, non infectious inflammation or uncontrollable systemic diseases (such as diabetes, hypertension, pulmonary fibrosis and acute pneumonia, etc.)
16. Known allergy to the study drug or any of its excipients, or severe allergic reactions to other monoclonal antibodies
17. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS)
18. Untreated active hepatitis B was defined as HBV-DNA ≥ 500 IU / ml;Hepatitis C, defined as HCV-RNA higher than the detection limit of the analytical method;Or combined with hepatitis B and C co infection
19. In the first 6 months, the following conditions occurred: myocardial infarction, severe / unstable angina pectoris, New York Heart Association （NYHA ）grade 2 or above cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmias, and symptomatic congestive heart failure
20. Hypertension was poorly controlled by drug therapy (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg)
21. Systemic use of antibiotics for more than 7 days in 4 weeks before randomization, or fever of unknown origin > 38.5 ° C during screening period / before first administration (fever due to tumor can be included in the group according to the judgment of the researcher)
22. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
23. Participated in any other drug clinical study within 4 weeks before randomization, or no more than 5 half-life from the last study
24. A history of psychotropic substance abuse or abuse is known
25. The presence of other laboratory abnormalities with severe physical or mental illness may increase the risk of participating in the study, or interfere with the results of the study and patients considered unsuitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
the appropriate dose of Bevacizumab | 1.5-3months
  According to the incidence of dose-limited toxic dose -limiting toxicity (DLT) after 2 and 4 cycles of Ib phase treatment, the appropriate dose of Bevacizumab combination was determined.
the objective Response Rate (ORR) of the experimental group. | 2years
  The main purpose of phase II is the objective Response Rate (ORR) of the experimental group.

SECONDARY OUTCOMES:
progression-free survival（PFS） | 1-2years
  Refers to the time between the patient's admission to the treatment and the disease progression
overall survival (OS) | 1-3years
  Refers to the time from admission to treatment to death of patients
disease control rate (DCR) | 1-3years
  Refers to the proportion of people who receive this program in the whole patient population and achieve complete response ,partial response or stable disease and last for a period of time

CONTACTS AND LOCATIONS:
Overall Officials: Liu Ming, Professor, Study Chair — West China Hospital
Locations (1):
- Liu Ming, Chengdu, China

REFERENCES:
- [Background] Van Cutsem E, de Haas S, Kang YK, Ohtsu A, Tebbutt NC, Ming Xu J, Peng Yong W, Langer B, Delmar P, Scherer SJ, Shah MA. Bevacizumab in combination with chemotherapy as first-line therapy in advanced gastric cancer: a biomarker evaluation from the AVAGAST randomized phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2119-27. doi: 10.1200/JCO.2011.39.9824. Epub 2012 May 7. PMID 22565005
- [Background] Han K, Jin J, Maia M, Lowe J, Sersch MA, Allison DE. Lower exposure and faster clearance of bevacizumab in gastric cancer and the impact of patient variables: analysis of individual data from AVAGAST phase III trial. AAPS J. 2014 Sep;16(5):1056-63. doi: 10.1208/s12248-014-9631-6. Epub 2014 Jun 19. PMID 24942210
- [Background] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- [Background] Kang YK, Chen LT, Ryu MH, Oh DY, Oh SC, Chung HC, Lee KW, Omori T, Shitara K, Sakuramoto S, Chung IJ, Yamaguchi K, Kato K, Sym SJ, Kadowaki S, Tsuji K, Chen JS, Bai LY, Oh SY, Choda Y, Yasui H, Takeuchi K, Hirashima Y, Hagihara S, Boku N. Nivolumab plus chemotherapy versus placebo plus chemotherapy in patients with HER2-negative, untreated, unresectable advanced or recurrent gastric or gastro-oesophageal junction cancer (ATTRACTION-4): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):234-247. doi: 10.1016/S1470-2045(21)00692-6. Epub 2022 Jan 11. PMID 35030335
- [Background] Shitara K, Van Cutsem E, Bang YJ, Fuchs C, Wyrwicz L, Lee KW, Kudaba I, Garrido M, Chung HC, Lee J, Castro HR, Mansoor W, Braghiroli MI, Karaseva N, Caglevic C, Villanueva L, Goekkurt E, Satake H, Enzinger P, Alsina M, Benson A, Chao J, Ko AH, Wainberg ZA, Kher U, Shah S, Kang SP, Tabernero J. Efficacy and Safety of Pembrolizumab or Pembrolizumab Plus Chemotherapy vs Chemotherapy Alone for Patients With First-line, Advanced Gastric Cancer: The KEYNOTE-062 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1571-1580. doi: 10.1001/jamaoncol.2020.3370. PMID 32880601
- [Background] Fukumura D, Kloepper J, Amoozgar Z, Duda DG, Jain RK. Enhancing cancer immunotherapy using antiangiogenics: opportunities and challenges. Nat Rev Clin Oncol. 2018 May;15(5):325-340. doi: 10.1038/nrclinonc.2018.29. Epub 2018 Mar 6. PMID 29508855
- [Background] Lee MS, Ryoo BY, Hsu CH, Numata K, Stein S, Verret W, Hack SP, Spahn J, Liu B, Abdullah H, Wang Y, He AR, Lee KH; GO30140 investigators. Atezolizumab with or without bevacizumab in unresectable hepatocellular carcinoma (GO30140): an open-label, multicentre, phase 1b study. Lancet Oncol. 2020 Jun;21(6):808-820. doi: 10.1016/S1470-2045(20)30156-X. PMID 32502443
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Ren Z, Xu J, Bai Y, Xu A, Cang S, Du C, Li Q, Lu Y, Chen Y, Guo Y, Chen Z, Liu B, Jia W, Wu J, Wang J, Shao G, Zhang B, Shan Y, Meng Z, Wu J, Gu S, Yang W, Liu C, Shi X, Gao Z, Yin T, Cui J, Huang M, Xing B, Mao Y, Teng G, Qin Y, Wang J, Xia F, Yin G, Yang Y, Chen M, Wang Y, Zhou H, Fan J; ORIENT-32 study group. Sintilimab plus a bevacizumab biosimilar (IBI305) versus sorafenib in unresectable hepatocellular carcinoma (ORIENT-32): a randomised, open-label, phase 2-3 study. Lancet Oncol. 2021 Jul;22(7):977-990. doi: 10.1016/S1470-2045(21)00252-7. Epub 2021 Jun 15. PMID 34143971
- [Background] Rini BI, Powles T, Atkins MB, Escudier B, McDermott DF, Suarez C, Bracarda S, Stadler WM, Donskov F, Lee JL, Hawkins R, Ravaud A, Alekseev B, Staehler M, Uemura M, De Giorgi U, Mellado B, Porta C, Melichar B, Gurney H, Bedke J, Choueiri TK, Parnis F, Khaznadar T, Thobhani A, Li S, Piault-Louis E, Frantz G, Huseni M, Schiff C, Green MC, Motzer RJ; IMmotion151 Study Group. Atezolizumab plus bevacizumab versus sunitinib in patients with previously untreated metastatic renal cell carcinoma (IMmotion151): a multicentre, open-label, phase 3, randomised controlled trial. Lancet. 2019 Jun 15;393(10189):2404-2415. doi: 10.1016/S0140-6736(19)30723-8. Epub 2019 May 9. PMID 31079938
- [Background] Socinski MA, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kelsch C, Lee A, Coleman S, Deng Y, Shen Y, Kowanetz M, Lopez-Chavez A, Sandler A, Reck M; IMpower150 Study Group. Atezolizumab for First-Line Treatment of Metastatic Nonsquamous NSCLC. N Engl J Med. 2018 Jun 14;378(24):2288-2301. doi: 10.1056/NEJMoa1716948. Epub 2018 Jun 4. PMID 29863955
- [Background] Sugawara S, Lee JS, Kang JH, Kim HR, Inui N, Hida T, Lee KH, Yoshida T, Tanaka H, Yang CT, Nishio M, Ohe Y, Tamura T, Yamamoto N, Yu CJ, Akamatsu H, Namba Y, Sumiyoshi N, Nakagawa K. Nivolumab with carboplatin, paclitaxel, and bevacizumab for first-line treatment of advanced nonsquamous non-small-cell lung cancer. Ann Oncol. 2021 Sep;32(9):1137-1147. doi: 10.1016/j.annonc.2021.06.004. Epub 2021 Jun 15. PMID 34139272
- [Background] Colombo N, Dubot C, Lorusso D, Caceres MV, Hasegawa K, Shapira-Frommer R, Tewari KS, Salman P, Hoyos Usta E, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Toker S, Li K, Keefe SM, Monk BJ; KEYNOTE-826 Investigators. Pembrolizumab for Persistent, Recurrent, or Metastatic Cervical Cancer. N Engl J Med. 2021 Nov 11;385(20):1856-1867. doi: 10.1056/NEJMoa2112435. Epub 2021 Sep 18. PMID 34534429
- [Background] Antoniotti C, Rossini D, Pietrantonio F, Catteau A, Salvatore L, Lonardi S, Boquet I, Tamberi S, Marmorino F, Moretto R, Ambrosini M, Tamburini E, Tortora G, Passardi A, Bergamo F, Kassambara A, Sbarrato T, Morano F, Ritorto G, Borelli B, Boccaccino A, Conca V, Giordano M, Ugolini C, Fieschi J, Papadopulos A, Massoue C, Aprile G, Antonuzzo L, Gelsomino F, Martinelli E, Pella N, Masi G, Fontanini G, Boni L, Galon J, Cremolini C; GONO Foundation Investigators. Upfront FOLFOXIRI plus bevacizumab with or without atezolizumab in the treatment of patients with metastatic colorectal cancer (AtezoTRIBE): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2022 Jul;23(7):876-887. doi: 10.1016/S1470-2045(22)00274-1. Epub 2022 May 27. PMID 35636444
- [Result] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Result] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Result] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Result] Fuchs CS, Shitara K, Di Bartolomeo M, Lonardi S, Al-Batran SE, Van Cutsem E, Ilson DH, Alsina M, Chau I, Lacy J, Ducreux M, Mendez GA, Alavez AM, Takahari D, Mansoor W, Enzinger PC, Gorbounova V, Wainberg ZA, Hegewisch-Becker S, Ferry D, Lin J, Carlesi R, Das M, Shah MA; RAINFALL Study Group. Ramucirumab with cisplatin and fluoropyrimidine as first-line therapy in patients with metastatic gastric or junctional adenocarcinoma (RAINFALL): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):420-435. doi: 10.1016/S1470-2045(18)30791-5. Epub 2019 Feb 1. PMID 30718072
- [Result] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Derived] Dai R, Zhang P, Cheng M, Bi F, Zhou J, Liu M. CapeOX (capecitabine and oxaliplatin) combined with sintilimab and bevacizumab biosimilar (IBI305) for first-line treatment of advanced gastric or oesophagogastric junction adenocarcinoma: study protocol for a single-arm, phase Ib/II trial. BMJ Open. 2026 Jan 9;16(1):e086005. doi: 10.1136/bmjopen-2024-086005. PMID 41513419
- See also: ESMO — https://www.esmo.org/content/search?searchText=Sintilimab+plus+chemotherapy+%28chemo%29+versus+chemo+as+first-line+treatment+for+advanced+gastric+or+gastroesophageal+junction+%28G%2FGEJ%29+adenocarcino+%28ORIENT-16%29%3A+First+results+of+a+randomized%2C+double-blind%2C+phase+III+study.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT05640609/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT05640609/ICF_001.pdf